CLINICAL TRIAL: NCT06314958
Title: Predicting Recurrence-Free Survival in Stage III and High-Risk Stage II Colorectal Cancer After Curative-Intent Treatment
Brief Title: Stage II/III Colorectal Cancer Recurrence
Acronym: CENSURE
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/CENSURE
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma; Colorectal Cancer Stage II; Colorectal Cancer Stage III; Colorectal Cancer Recurrent
Keywords: Recurrence-free Survival (RFS); Overall Survival (OS); Methylation; DNA methylation; carcinoembryonic antigen (CEA)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-fixed and paraffin-embedded samples derived from the primary tumor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stage II/III Colorectal Cancer, with Recurrence (Training): Stage II/III Colorectal Cancer patients who received treatment with surgery and adjuvant chemotherapy, and experienced recurrence within five years.
  Interventions: Other: CENSURE
- Stage II/III Colorectal Cancer, without Recurrence (Training): Stage II/III Colorectal Cancer patients who received treatment with surgery and adjuvant chemotherapy, and did not experience recurrence within five years.
  Interventions: Other: CENSURE
- Stage II/III Colorectal Cancer, with Recurrence (Validation): Stage II/III Colorectal Cancer patients who received treatment with surgery and adjuvant chemotherapy, and experienced recurrence within five years.
  Interventions: Other: CENSURE
- Stage II/III Colorectal Cancer, without Recurrence (Validation): Stage II/III Colorectal Cancer patients who received treatment with surgery and adjuvant chemotherapy, and did not experience recurrence within five years.
  Interventions: Other: CENSURE

INTERVENTIONS:
Other: CENSURE — A panel of CpG sites, whose methylation level is tested in macro-dissected formalin-fixed and paraffin-embedded (FFPE) samples derived from the primary tumor.
  Other Names: CENSURE (CpG mEthylation-based epigeNetic SignatURE)

SUMMARY:
This study will develop an assay to predict disease recurrence in patients with stage II/III CRC after receiving adjuvant chemotherapy, using genome-wide DNA methylation.

DETAILED DESCRIPTION:
Adjuvant chemotherapy (ACT) is the standard clinical care for patients with stage III or high-risk stage II colorectal cancer (CRC) after curative-intent resection. Nonetheless, more than 30% of patients experience CRC recurrence. Accurate prediction of recurrence risk in stage II/III CRC patients who undergo ACT is crucial for determining the necessity and duration of ACT, as well as for tailoring novel treatment strategies for these patients.

This study will comprise three phases

1. A systematic and comprehensive CpG methylation-based epigenetic biomarker discovery phase to identify the differentially methylated CpG sites associated with recurrence-free survival (RFS) < 5 years and > 5 years. In this phase, LASSO-based machine learning algorithms will be used to optimize the biomarker candidates.
2. A tissue-based clinical assay development phase by quantitative pyrosequencing
3. An independent validation phase.

At completion, this study will validate a tissue-based assay to predict the development of recurrence after the completion of chemotherapy in patients with stage III and II CRC

ELIGIBILITY:
Inclusion Criteria:

* Stage II (high-risk) or III colorectal cancer (TNM classification, 8th edition).
* Received standard diagnostic, staging, and therapeutic procedures as per local guidelines
* Received stage-specific curative-intent resection followed by adjuvant chemotherapy.
* Confirmed cancer-free survivorship confirmed at the time of study inclusion.

Exclusion Criteria:

* Lack of written informed consent.
* Development of recurrence in the first 6 months following adjuvant chemotherapy completion.
* Hereditary colorectal cancer syndromes (identified through genetic testing)
* Inflammatory bowel diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two independent cohorts of colorectal cancer survivors (high-risk stage II and stage III), who received curative-intent surgery and adjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival | Up to 120 months
  Time from treatment completion to development of recurrence (or death)

SECONDARY OUTCOMES:
Overall Survival | Up to 120 months
  Time from treatment completion to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (4):
- City of Hope Medical Center, Monrovia, California, United States
- Second Affiliated Hospital of Dalian Medical University, Dalian, China
- Spain (2):
  - Barcelona University, Barcelona
  - La Paz University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Frei AL, McGuigan A, Sinha RRAK, Jabbar F, Gneo L, Tomasevic T, Harkin A, Iveson T, Saunders MP, Oien KA, Maka N, Pezzella F, Campo L, Browne M, Glaire M, Kildal W, Danielsen HE, Hay J, Edwards J, Sansom O, Kelly C, Tomlinson I, Kerr R, Kerr D, Domingo E; TransSCOT consortium; Church DN, Koelzer VH. Multiplex analysis of intratumoural immune infiltrate and prognosis in patients with stage II-III colorectal cancer from the SCOT and QUASAR 2 trials: a retrospective analysis. Lancet Oncol. 2024 Feb;25(2):198-211. doi: 10.1016/S1470-2045(23)00560-0. PMID 38301689
- [Background] Argiles G, Tabernero J, Labianca R, Hochhauser D, Salazar R, Iveson T, Laurent-Puig P, Quirke P, Yoshino T, Taieb J, Martinelli E, Arnold D; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Localised colon cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Oct;31(10):1291-1305. doi: 10.1016/j.annonc.2020.06.022. Epub 2020 Jul 20. No abstract available. PMID 32702383
- [Background] Liu Z, Guo C, Dang Q, Wang L, Liu L, Weng S, Xu H, Lu T, Sun Z, Han X. Integrative analysis from multi-center studies identities a consensus machine learning-derived lncRNA signature for stage II/III colorectal cancer. EBioMedicine. 2022 Jan;75:103750. doi: 10.1016/j.ebiom.2021.103750. Epub 2021 Dec 15. PMID 34922323
- [Background] Feng Q, Chang W, Mao Y, He G, Zheng P, Tang W, Wei Y, Ren L, Zhu D, Ji M, Tu Y, Qin X, Xu J. Tumor-associated Macrophages as Prognostic and Predictive Biomarkers for Postoperative Adjuvant Chemotherapy in Patients with Stage II Colon Cancer. Clin Cancer Res. 2019 Jul 1;25(13):3896-3907. doi: 10.1158/1078-0432.CCR-18-2076. Epub 2019 Apr 15. PMID 30988081
- [Background] Osterman E, Glimelius B. Recurrence Risk After Up-to-Date Colon Cancer Staging, Surgery, and Pathology: Analysis of the Entire Swedish Population. Dis Colon Rectum. 2018 Sep;61(9):1016-1025. doi: 10.1097/DCR.0000000000001158. PMID 30086050
- [Background] Varghese A. Chemotherapy for Stage II Colon Cancer. Clin Colon Rectal Surg. 2015 Dec;28(4):256-61. doi: 10.1055/s-0035-1564430. PMID 26648796
- [Background] Bockelman C, Engelmann BE, Kaprio T, Hansen TF, Glimelius B. Risk of recurrence in patients with colon cancer stage II and III: a systematic review and meta-analysis of recent literature. Acta Oncol. 2015 Jan;54(1):5-16. doi: 10.3109/0284186X.2014.975839. Epub 2014 Nov 28. PMID 25430983
- [Background] Cheng E, Ou FS, Ma C, Spiegelman D, Zhang S, Zhou X, Bainter TM, Saltz LB, Niedzwiecki D, Mayer RJ, Whittom R, Hantel A, Benson A, Atienza D, Messino M, Kindler H, Giovannucci EL, Van Blarigan EL, Brown JC, Ng K, Gross CP, Meyerhardt JA, Fuchs CS. Diet- and Lifestyle-Based Prediction Models to Estimate Cancer Recurrence and Death in Patients With Stage III Colon Cancer (CALGB 89803/Alliance). J Clin Oncol. 2022 Mar 1;40(7):740-751. doi: 10.1200/JCO.21.01784. Epub 2022 Jan 7. PMID 34995084
- [Background] Dienstmann R, Mason MJ, Sinicrope FA, Phipps AI, Tejpar S, Nesbakken A, Danielsen SA, Sveen A, Buchanan DD, Clendenning M, Rosty C, Bot B, Alberts SR, Milburn Jessup J, Lothe RA, Delorenzi M, Newcomb PA, Sargent D, Guinney J. Prediction of overall survival in stage II and III colon cancer beyond TNM system: a retrospective, pooled biomarker study. Ann Oncol. 2017 May 1;28(5):1023-1031. doi: 10.1093/annonc/mdx052. PMID 28453697
- [Background] Konishi T, Shimada Y, Hsu M, Tufts L, Jimenez-Rodriguez R, Cercek A, Yaeger R, Saltz L, Smith JJ, Nash GM, Guillem JG, Paty PB, Garcia-Aguilar J, Gonen M, Weiser MR. Association of Preoperative and Postoperative Serum Carcinoembryonic Antigen and Colon Cancer Outcome. JAMA Oncol. 2018 Mar 1;4(3):309-315. doi: 10.1001/jamaoncol.2017.4420. PMID 29270608
- [Background] Nicholson BD, Shinkins B, Pathiraja I, Roberts NW, James TJ, Mallett S, Perera R, Primrose JN, Mant D. Blood CEA levels for detecting recurrent colorectal cancer. Cochrane Database Syst Rev. 2015 Dec 10;2015(12):CD011134. doi: 10.1002/14651858.CD011134.pub2. PMID 26661580
- [Background] Dienstmann R, Villacampa G, Sveen A, Mason MJ, Niedzwiecki D, Nesbakken A, Moreno V, Warren RS, Lothe RA, Guinney J. Relative contribution of clinicopathological variables, genomic markers, transcriptomic subtyping and microenvironment features for outcome prediction in stage II/III colorectal cancer. Ann Oncol. 2019 Oct 1;30(10):1622-1629. doi: 10.1093/annonc/mdz287. PMID 31504112
- [Background] Hutchins G, Southward K, Handley K, Magill L, Beaumont C, Stahlschmidt J, Richman S, Chambers P, Seymour M, Kerr D, Gray R, Quirke P. Value of mismatch repair, KRAS, and BRAF mutations in predicting recurrence and benefits from chemotherapy in colorectal cancer. J Clin Oncol. 2011 Apr 1;29(10):1261-70. doi: 10.1200/JCO.2010.30.1366. Epub 2011 Mar 7. PMID 21383284
- [Background] Pages F, Mlecnik B, Marliot F, Bindea G, Ou FS, Bifulco C, Lugli A, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert C, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang JY, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Angelova M, Vasaturo A, Maby P, Church SE, Angell HK, Lafontaine L, Bruni D, El Sissy C, Haicheur N, Kirilovsky A, Berger A, Lagorce C, Meyers JP, Paustian C, Feng Z, Ballesteros-Merino C, Dijkstra J, van de Water C, van Lent-van Vliet S, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Itoh K, Patel PS, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Sargent DJ, Fox BA, Galon J. International validation of the consensus Immunoscore for the classification of colon cancer: a prognostic and accuracy study. Lancet. 2018 May 26;391(10135):2128-2139. doi: 10.1016/S0140-6736(18)30789-X. Epub 2018 May 10. PMID 29754777
- [Background] Yothers G, O'Connell MJ, Lee M, Lopatin M, Clark-Langone KM, Millward C, Paik S, Sharif S, Shak S, Wolmark N. Validation of the 12-gene colon cancer recurrence score in NSABP C-07 as a predictor of recurrence in patients with stage II and III colon cancer treated with fluorouracil and leucovorin (FU/LV) and FU/LV plus oxaliplatin. J Clin Oncol. 2013 Dec 20;31(36):4512-9. doi: 10.1200/JCO.2012.47.3116. Epub 2013 Nov 12. PMID 24220557
- [Background] Henriksen TV, Tarazona N, Frydendahl A, Reinert T, Gimeno-Valiente F, Carbonell-Asins JA, Sharma S, Renner D, Hafez D, Roda D, Huerta M, Rosello S, Madsen AH, Love US, Andersen PV, Thorlacius-Ussing O, Iversen LH, Gotschalck KA, Sethi H, Aleshin A, Cervantes A, Andersen CL. Circulating Tumor DNA in Stage III Colorectal Cancer, beyond Minimal Residual Disease Detection, toward Assessment of Adjuvant Therapy Efficacy and Clinical Behavior of Recurrences. Clin Cancer Res. 2022 Feb 1;28(3):507-517. doi: 10.1158/1078-0432.CCR-21-2404. Epub 2021 Oct 8. PMID 34625408
- [Background] Romesser PB, Sanchez-Vega F, Joshua Smith J. A methylation-based prognostic signature in stage II colorectal patients: Considerations for clinical adoption. J Natl Cancer Inst. 2023 Jan 10;115(1):8-11. doi: 10.1093/jnci/djac184. No abstract available. PMID 36171662